CLINICAL TRIAL: NCT02117388
Title: Treatments for Insomnia: Mediators, Moderators and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jerome Yesavage, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27264; 1R01MH101468-01 (NIH)
Record Dates: First submitted 2014-02-04; First posted 2014-04-17 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Insomnia
Keywords: Older adults; insomnia; CBT-I (cognitive behavioral therapy-insomnia); Behavioral Therapy; SRT (sleep restriction therapy); Cognitive Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Psychotherapy, Multiple

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy is designed to identify incorrect ideas about sleep, challenge their validity, and replace them with correct information. This therapy tries to reduce worry, anxiety, and fear that one won't sleep by providing accurate information about sleep.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Sleep Restriction (Experimental): Sleep Restriction therapy will limit the time participants spend in bed in order to make sure they are sleepy enough to fall asleep quickly.
  Interventions: Behavioral: Sleep Restriction
- Combined Therapy Treatment for Insomnia (Experimental): Combined Therapy involves combining Sleep Restriction and Cognitive Therapy so that the two therapies reinforce each other.
  Interventions: Behavioral: Combined Therapy

INTERVENTIONS:
Behavioral: Sleep Restriction — Sleep Restriction therapy will limit the time spent in bed in order to make sure participants are sleepy enough to fall asleep quickly.
  Arms: Sleep Restriction
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy is designed to identify incorrect ideas about sleep, challenge their validity, and replace them with correct information. This therapy tries to reduce worry, anxiety, and fear that one won't sleep by providing accurate information about sleep.
  Arms: Cognitive Behavioral Therapy
Behavioral: Combined Therapy — Sleep Restriction and Cognitive Therapy will be combined so that the two therapies reinforce each other.
  Arms: Combined Therapy Treatment for Insomnia

SUMMARY:
The purpose of this study is to evaluate the relative efficacy and effectiveness of specific components of cognitive behavioral therapies for insomnia: sleep restriction (SR) and cognitive therapy (CT) in comparison to combined SR and CT (SR+CT).

DETAILED DESCRIPTION:
As many as one in three older adults may experience insomnia. Older adults are the most frequent users of hypnotic medications. Although safer, use of even the latest "sleeping pills" can lead to cognitive impairment and risk of falls. Thus, it is not surprising that non-pharmacological treatments for insomnia have been pursued as alternatives to medications, with some suggesting they should be the "first line of therapy". We propose a randomized clinical trial to evaluate the relative efficacy and effectiveness of specific components of cognitive behavioral therapies for insomnia (CBT-I): sleep restriction (SR) and cognitive therapy (CT) in comparison to combined SR and CT (SR+CT). We hypothesize that because the proposed mechanisms of action of CT versus SR substantially differ, their combination may have additive effects. Even though the mechanisms of action of SR and CT may differ, no data exists to document that the addition of one to the other provides more overall clinical benefit than either intervention alone. Finally, to better understand "how" and "in whom" SR and CT work, we plan to formally evaluate selected mediators and moderators of the clinical effect including physiological measures of anxiety and arousal. Three treatments (SR, CT, and SR+CT) will be compared in a randomized clinical trial with a parallel groups design. Efficacy and effectiveness data will be collected prior to the beginning of treatment, after 6 weeks of treatment, and at the end of a 6-month follow-up. These efforts follow the National Institute of Mental Health Strategic Plan Strategy 3.1 to develop innovative interventions and designs for intervention studies, in this case, to promote a new intervention trial that focuses on the mediators and moderators of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of any racial or ethnic group, aged 60 years old or older
* Independent living (not in nursing home, etc.)
* English-speaking
* Subjective complaint of insomnia associated with daytime impairment or distress
* DSM 5 (Diagnostic and Statistical Manual V) diagnosis of insomnia
* Score >10 on the Insomnia Severity Indexa
* Must live within 40 miles of Stanford University

Exclusion Criteria:

* Montreal Cognitive Assessment Scale <20
* Apnea-hypopnea index >10 or Periodic limb movement associated arousals > 5 per hour
* Use of medication specifically prescribed for sleep and unwilling or unable to discontinue > one week prior to baseline data collection.
* Acute or unstable chronic illness: including but not limited to insulin dependent diabetes (adult onset diabetes, controlled with oral medications or diet is acceptable); uncontrolled thyroid disease, kidney, prostate or bladder conditions causing excessively frequent urination (> 3 times per night); medically unstable congestive heart failure, angina, other severe cardiac illness as defined by treatment regimen changes in the prior 3 months; stroke with serious sequelae; cancer if < 1 year since end of treatment; asthma, emphysema, or other severe respiratory diseases uncontrolled with medications; conditions associated with chronic pain such as fibromyalgia; and neurological disorders such as Alzheimer's disease, Parkinson's disease and unstable epilepsy as defined by treatment regimen changes in the prior 3 months.
* Use of CNS (central nervous system) active medications that would significantly impact sleep or alertness is allowed as long as the dose, timing, and formulation are stable (> 4 weeks).
* Excessive caffeine consumption (≥ three cups per day), excessive alcohol consumption (> 14 drinks per week or > 4 drinks per occasion), or illicit substances (by self-report).
* Major psychiatric diagnosis on Axis I of DSM-IV as tested by the Mini International Neuropsychiatric Interview (Version 5.0).
* Lives more than 40 miles from Stanford University

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Screening, End of 6-week treatment, 6-month follow-up
  Subject's subjective evaluation of their sleep.

SECONDARY OUTCOMES:
Cognitive Arousal | Screening, end of 6-week treatment, 6-month followup
  Score on Penn State Worry Questionnaire, and Dysfunctional Beliefs and Attitudes about Sleep Scale.
  Both measures have been found to be successful in measuring mediators and moderators of treatment response.
Chronic Stress | Screening, end of 6-week treatment, 6-month followup
  We are using two of the most widely utilized psychometric indices of past, present and chronic stress exposure: 1) the Trauma History Questionnaire, and 2) the Life Stressor Checklist revised, a clinical interview for lifetime exposure to stressful life events.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome A. Yesavage, MD, Principal Investigator — VA/Stanford
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] O'Hora KP, Morehouse AB, Freidman L, Posner D, Ahmadi M, Hernandez B, Burda KF, Kushida C, Zeitzer JM, Lazzeroni LC, Manber R, Yesavage J, Goldstein-Piekarski AN. Comparative effectiveness and predictors of cognitive behavioral therapy for insomnia and its components in older adults: main outcomes of a randomized dismantling trial. J Clin Sleep Med. 2025 Oct 1;21(10):1679-1695. doi: 10.5664/jcsm.11756. PMID 40476601